CLINICAL TRIAL: NCT04473690
Title: A Phase I/II, First-in-human, Observer-blinded, Randomized, Placebo-controlled, Parallel Group Study to Evaluate the Safety and Immunogenicity of TAP-COVID-19 SARS-CoV-2 Vaccine With CpG Adjuvant in Healthy Adults Aged 18-49 and 50-85
Brief Title: KBP-201 COVID-19 Vaccine Trial in Healthy Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: KBio Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KBP-201
Record Dates: First submitted 2020-07-14; First posted 2020-07-16 (Actual); Results first posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Covid19
Keywords: Vaccine; Covid19 Vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose KBP-COVID-19 and adjuvant (Experimental): Two age groups.
  Part A (18-49 years).
  Part B (50-85 years).
  All subjects in these groups will receive the low dose of KBP-COVID-19
  Interventions: Biological: Low Dose of KBP-COVID-19
- High Dose KBP-COVID-19 and adjuvant (Experimental): Two age groups.
  Part A (18-49 years).
  Part B (50-85 years).
  All subjects in these groups will receive the high dose of KBP-COVID-19
  Interventions: Biological: High Dose of KBP-COVID-19
- Placebo (Placebo Comparator): Two age groups.
  Part A (18-49 years).
  Part B (50-85 years).
  All subjects in these groups will receive placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Low Dose of KBP-COVID-19 — Low Dose of KBP-COVID-19 and adjuvant
  Arms: Low Dose KBP-COVID-19 and adjuvant
Biological: High Dose of KBP-COVID-19 — High Dose of KBP-COVID-19 and adjuvant
  Arms: High Dose KBP-COVID-19 and adjuvant
Biological: Placebo — Buffered saline solution
  Arms: Placebo

SUMMARY:
This is an First In Human (FIH), observer-blinded, randomized, placebo-controlled, parallel group study to evaluate the safety and immunogenicity of KBP-COVID-19 plus CPG adjuvant vaccine in healthy adult subjects in 2 age groups, Part A (18-49 years) and Part B (50-85 years).

DETAILED DESCRIPTION:
Subjects will be screened up to 14 days (Day -14 to Day -1) before randomization.

Approximately 90 eligible healthy adults ages 18-49 years (inclusive) will be enrolled for Part A and 90 eligible healthy seronegative adults ages 50-85 years will be enrolled for Part B.

Sentinel dosing (three subjects in each group) will be utilized in this FIH study. Sentinel cohorts will be used for the following groups:

Part A (18-49 years) low dose Part B (50-85 years) low dose Part A (18-49 years) high dose Part B (50-85 years) high dose

Overall, subjects will be randomized in a 1:1:1 ratio to receive study vaccine or placebo by IM injection on Days 1 and 22.

All study visits will be conducted at the clinical sites on an outpatient basis. Subjects will participate in the study for approximately 1 year from the first dose.

ELIGIBILITY:
Inclusion Criteria:

1. Subject read, understood, and signed the informed consent form (ICF).
2. Healthy adult males and females 18-49 years of age (Part A) or 50-85 years of age (Part B), inclusive, at screening.
3. RT-PCR negative at time of screening.
4. Body mass index (BMI) of ≥ 18 and ≤ 30 kg/m2 at screening. BMI = weight (kg)/(height [m])2.
5. Must be in general good health before study participation with no clinically relevant abnormalities that could interfere with study assessments.
6. Women of childbearing potential (WOCBP) and men whose sexual partners are WOCBP must be able and willing to use at least 1 highly effective method of contraception (ie, include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy, hormonal oral [in combination with male condoms with spermicide], transdermal, implant, or injection, barrier [ie, condom, diaphragm with spermicide]; intrauterine device; vasectomized partner [6 months minimum], clinically sterile partner; or abstinence) during the study. A female subject is considered to be a WOCBP after menarche and until she is in a postmenopausal state for 12 consecutive months (without an alternative medical cause) or otherwise permanently sterile. Note: Subjects not of childbearing potential are not required to use any other forms of contraception during the study. Non-childbearing potential is defined as subject confirmed:

   * Surgical sterilization (eg, bilateral oophorectomy, bilateral salpingectomy, bilateral occlusion by cautery [Essure System is not acceptable], hysterectomy, or tubal ligation).
   * Postmenopausal (defined as permanent cessation of menstruation for at least 12 consecutive months prior to screening) with FSH ≥ 30 mIU/mL at screening.
7. WOCBP must have a negative urine pregnancy test before each vaccination.
8. Must be able to attend all visits, including unscheduled visits if respiratory symptoms develop during the study, for the duration of the study and comply with all study procedures, including daily completion of the Diary Card for 7 days after each injection.

Exclusion Criteria

1. History of an acute or chronic medical condition including dementia that, in the opinion of the Investigator, would render vaccination unsafe or would interfere with the evaluation of responses. Chronic conditions that are NOT included on the Center for Disease Control's list of subjects at higher risk for severe illness from SARS-CoV-2 are acceptable if the condition has been stable for the 3 months prior to vaccine administration (Day 1), with no medication changes, and no hospitalization in the past 6 months.
2. History of any medical conditions that place subjects at higher risk for severe illness due to SARS-CoV-2 including but not limited to cancer, chronic kidney disease at any stage, chronic lung disease, dementia or other neurological conditions, diabetes (Type 1 or Type 2), Down syndrome, heart conditions, human immunodeficiency virus (HIV) infection, immunocompromised state (weakened immune system), liver disease, overweight/obesity, pregnancy, sickle cell disease or thalassemia, smoker (current or former), transplants (solid organ or blood stem cell), stroke or cerebrovascular disease, and substance use disorders.
3. History of ongoing clinical condition or medication or treatments that may adversely affect the immune system.
4. Individuals who are PCR positive for SARS-CoV-2 at screening or prior to second dose of TAP-COVID-19 vaccine.
5. Individuals who are at increased risk of exposure to SARS-CoV-2 (eg, healthcare workers, emergency responders).
6. Close contact of anyone known to have SARS-CoV-2 infection within 30 days prior to vaccine administration.
7. Living in a group care facility (eg, assisted living or nursing home).
8. Individuals with any elevated (Grade 1 or higher) laboratory test assessed as clinically significant for age by the Investigator at screening.
9. Individuals with any elevated (Grade 1 or higher) liver function enzyme at screening,
10. Active neoplastic disease (excluding nonmelanoma skin cancer that was successfully treated) or a history of any hematological malignancy. "Active" is defined as having received treatment within the past 5 years.
11. Long-term (greater than 2 weeks) use of oral or parenteral steroids, high-dose inhaled steroids (>800 μg/day of beclomethasone dipropionate or equivalent), or immunomodulatory drugs within 6 months before screening (nasal and topical steroids are allowed).
12. History of autoimmune, inflammatory disease, or potential immune-mediated medical conditions (Appendix B).
13. Women currently pregnant, lactating, or planning a pregnancy between enrollment and 181 days after randomization.
14. History of Guillain-Barré Syndrome.
15. History of anaphylactic-type reaction to injected vaccines.
16. Known or suspected hypersensitivity to 1 or more of the components of the vaccine, including thimerosal, tobacco, and CpG adjuvant.
17. History of alcohol abuse, illicit drug use, physical dependence to any opioid, or any history of drug abuse or addiction within 12 months of screening.
18. Acute illness or fever within 3 days before study enrollment (enrollment may be delayed for full recovery if acceptable to the Investigator).
19. Individuals currently participating or planning to participate in a study that involves an experimental agent (vaccine, drug, biologic, device, or medication); or who have received an experimental agent within 1 month (3 months for immunoglobulins) before enrollment in this study; or who expect to receive another experimental agent during participation in this study.
20. Receipt of immunoglobulin or another blood product within the 3 months before enrollment in this study or those who expect to receive immunoglobulin or another blood product during this study.
21. Individuals who intend to donate blood within 6 months after the first vaccination.
22. Individuals using prescription medications for prophylaxis of SARS-CoV-2.
23. Individuals who plan to receive another vaccine within the first 3 months of the study except influenza vaccine which should not be given within 2 weeks of study vaccine.
24. Receipt of any other approved SARS CoV 2 vaccine prior to the first study vaccine or within 90 days after administration of the first study vaccine.
25. Receipt of any other experimental coronavirus vaccine at any time prior to or during the study.
26. Receipt of any investigational vaccine or drug within 1 month of enrollment and through the end of the study (1 year after first vaccination).
27. Plan to travel outside the subjects' country of residence from enrollment through Day 43.
28. History of surgery or major trauma within 12 weeks of screening, or surgery planned during the study.
29. Significant blood loss (>450 mL) or has donated 1 or more units of blood or plasma within 6 weeks prior to study participation.
30. Strenuous activity (as assessed by the Investigator) within 48 hours prior to dosing (Days 1 and 22).
31. A positive urine drug screen without evidence of corresponding prescribed concomitant medication(s) at Screening.
32. Positive alcohol screen.
33. Positive screen for HIV-1 and HIV-2 antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibody.
34. Involved in the planning or conduct of this study.
35. Unwilling or unlikely to comply with the requirements of the study.
36. Subject is an employee, contractor, friend of or relative of any employee of Sponsor, contract research organization (CRO), study site or site affiliate.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Bratcher, Study Director — KBio Inc
Locations (8):
- United States (6):
  - Palm Beach Research Center, West Palm Beach, Florida
  - Velocity Clinical Research, Meridian, Idaho
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - PanAmerican Clinical Research, Brownsville, Texas
  - ICON, San Antonio, Texas
  - DM Clinical Research, Tomball, Texas
- Canada (2):
  - LMC Manna Research, Burlington, Burlington/Ontario
  - LMC Manna Research, Montreal, Point Claire, Quebec

IPD SHARING:
Plan to Share IPD: No
Plan is to share study data by dosing group in publications

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose KBP-COVID-19 and Adjuvant: Two age groups.
  Part A (18-49 years).
  Part B (50-85 years).
  All subjects in these groups will receive the low dose of KBP-COVID-19
  Low Dose of KBP-COVID-19: Low Dose of KBP-COVID-19 and adjuvant
- High Dose KBP-COVID-19 and Adjuvant: Two age groups.
  Part A (18-49 years).
  Part B (50-85 years).
  All subjects in these groups will receive the high dose of KBP-COVID-19
  High Dose of KBP-COVID-19: High Dose of KBP-COVID-19 and adjuvant
- Placebo: Two age groups.
  Part A (18-49 years).
  Part B (50-85 years).
  All subjects in these groups will receive placebo
  Placebo: Buffered saline solution
Period: Overall Study
Arm/Group | Low Dose KBP-COVID-19 and Adjuvant | High Dose KBP-COVID-19 and Adjuvant | Placebo
Started | 36 | 30 | 36
Completed | 31 | 28 | 32
Not Completed | 5 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose KBP-COVID-19 and Adjuvant | High Dose KBP-COVID-19 and Adjuvant | Placebo | Total
Number analyzed (Participants) | 36 | 30 | 36 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 36 | 30 | 35 | 101
  >=65 years | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 20 | 58
  Male | 15 | 13 | 16 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 2 | 4 | 4 | 10
  White | 33 | 24 | 31 | 88
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Solicited Administration Site Reactions
Description: Occurrence of Adverse Events
Time Frame: 7 days following the first vaccination on day 1 and 7 days following the second vaccination on day 22, up to 29 days
Population: number of subjects with solicited site reactions 7 day after two vaccinations
Measure: Number; unit: participants
Arm/Group | Low Dose KBP-COVID-19 and Adjuvant | High Dose KBP-COVID-19 and Adjuvant | Placebo
Number analyzed (Participants) | 34 | 29 | 35
participants | 19 | 15 | 20

2. Primary Outcome: Solicited Systemic Events
Description: Occurrence of Adverse Events
Time Frame: 7 days following the first vaccination on day 1 and 7 days following the second vaccination on day 22, up to 29 days
Population: Medically attended adverse reaction
Measure: Number; unit: Number of events
Arm/Group | Low Dose KBP-COVID-19 and Adjuvant | High Dose KBP-COVID-19 and Adjuvant | Placebo
Number analyzed (Participants) | 34 | 29 | 35
Number of events | 3 | 2 | 0

ADVERSE EVENTS:
Time Frame: From dosing to Day 43
Arm/Group | Low Dose KBP-COVID-19 and Adjuvant | High Dose KBP-COVID-19 and Adjuvant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/30 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/30 | 0/36
Other Adverse Events (participants affected / at risk) | 5/36 | 4/30 | 3/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose KBP-COVID-19 and Adjuvant (N=36) | High Dose KBP-COVID-19 and Adjuvant (N=30) | Placebo (N=36)
Injection site reactions (Investigations) | 5 (6) | 4 (5) | 3 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/90/NCT04473690/Prot_SAP_001.pdf